CLINICAL TRIAL: NCT05768022
Title: Origin to Insertion Kinesio Tapping vs Non-Directional Kinesio Tapping on Quadriceps Peak
Brief Title: Origin to Insertion Kinesio Tapping vs Non-Directional Kinesio Tapping on Quadriceps Peak Torque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Mohamed Moustafa Mohamed Ahmed, Assistant Professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 91177
Record Dates: First submitted 2023-02-18; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Quadriceps Muscle Atrophy

STUDY DESIGN:
Intervention Model Description: A Pretest posttest control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cura kinesio-taping (Experimental): 100 subjects (females and males) will receive kinesio taping from origin to insertion on the superficial muscles of Quadriceps femoris (VM,VL, RF).
  Interventions: Other: Cura Kensio-tapping
- Placebo (Placebo Comparator): 100 subjects (females and males) will receive placebo kinesio-taping across quadriceps.
  Interventions: Other: placebo

INTERVENTIONS:
Other: Cura Kensio-tapping — Cura tapes, a cotton strip with an acrylic adhesive. allows for unidirectional elasticity up to 60% beyond its resting length.
  Arms: Cura kinesio-taping
Other: placebo — placebo taping
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effect of kinesio tapping on electrical activity and peak torque of quadriceps during concentric and eccentric muscle contraction were carried out in the motion analysis Laboratory.

DETAILED DESCRIPTION:
A Pretest posttest control group design was used to. Two hundred normal subjects of both sexes were recruited.

Subjects were randomly assigned into two groups of equal number.

* Cura Kensio-tapping group: consisted of 100 subjects (females and males) will receive kinesio taping from origin to insertion on the superficial muscles of Quadriceps femoris (vastus medialis (VM), vastus lateralis (VL), rectus femoris (RF).
* Placebo-Group: consisted of 100 subjects (females and males) will receive placebo kinesio taping across quadriceps.

ELIGIBILITY:
Inclusion Criteria:

* Age must be ranged from 22-30 years.
* Body mass index must be ranged from 20-24.9 kg/m².

Exclusion Criteria:

* Knee or quadriceps disorders preventing physical stress.
* Cardiovascular or neurological problems.
* Athletic subjects.
* Smokers.
* Heavy caffeine intake subjects.

Ages: 22 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Peak Torque Measurement 1 | Before tapping.
  The peak torque of quadriceps muscle of dominant lower limb was measured using Biodex system 830-200 Isokinetic dynamometer.
Peak Torque Measurement 2 | After the application of tapping by 10 minutes
  The peak torque of quadriceps muscle of dominant lower limb was measured using Biodex system 830-200 Isokinetic dynamometer.
Peak Torque Measurement 3 | 24 hours after tapping.
  The peak torque of quadriceps muscle of dominant lower limb was measured using Biodex system 830-200 Isokinetic dynamometer.
Peak Torque Measurement 4 | 72 hours After tapping
  The peak torque of quadriceps muscle of dominant lower limb was measured using Biodex system 830-200 Isokinetic dynamometer.
Peak Torque Measurement 5 | 5 days after removal of tapping b
  The peak torque of quadriceps muscle of dominant lower limb was measured using Biodex system 830-200 Isokinetic dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Jizan, Gizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No